CLINICAL TRIAL: NCT01288313
Title: Effect of N-3 Polyunsaturated Fatty Acids Supplementation on the Human Milk Composition of Lactating Women: Nutritional Intervention With Rapeseed Oil and n-3 Margarine Compared to Standard Olive Oil
Brief Title: Effect of n-3 Polyunsaturated Fatty Acids Supplementation on Human Milk Composition of Lactating Women
Acronym: Oméga 3
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Collaborators: ITERG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 2010/35; 2008-058
Record Dates: First submitted 2011-01-31; First posted 2011-02-02 (Estimated); Last update posted 2014-08-20 (Estimated); Status verified 2014-08

CONDITIONS: Nursing Women
Keywords: human milk; polyunsaturated fatty acids; linolenic acid; rapeseed oil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- rapeseed oil (Experimental)
  Interventions: Dietary Supplement: nutritional intervention
- n-3 margarine and rapeseed oil (Experimental)
  Interventions: Dietary Supplement: nutritional intervention
- n-3 margarine (Experimental)
  Interventions: Dietary Supplement: nutritional intervention
- Olive oil (Active Comparator)
  Interventions: Dietary Supplement: nutritional intervention

INTERVENTIONS:
Dietary Supplement: nutritional intervention — Each diet will last 30 days. During the first period of 15 days, the mothers will receive mediterranean diet based on olive oil. Then, lactating women will receive 30gr/day rapeseed oil. Human milk will be collected during the first breastfeeding of the day (10 ml) at three times : Days 0 corresponding to the usual diet , at day 15 after the Mediterranean diet and at day 30, after the study diet.
  Arms: rapeseed oil
Dietary Supplement: nutritional intervention — Each diet will last 30 days. During the first period of 15 days, the mothers will receive mediterranean diet based on olive oil. Then, lactating women will receive diet associating 30gr/day of rapeseed oil and n-3 margarine. Human milk will be collected during the first breastfeeding of the day (10 ml) at three times : Days 0 corresponding to the usual diet , at day 15 after the Mediterranean diet and at day 30, after the study diet.
  Arms: n-3 margarine and rapeseed oil
Dietary Supplement: nutritional intervention — Each diet will last 30 days. During the first period of 15 days, the mothers will receive mediterranean diet based on olive oil. Then, lactating women will receive with 30gr/day n-3 margarine. Human milk will be collected during the first breastfeeding of the day (10 ml) at three times : Days 0 corresponding to the usual diet , at day 15 after the Mediterranean diet and at day 30, after the study diet.
  Arms: n-3 margarine
Dietary Supplement: nutritional intervention — Each diet will last 30 days. During the first period of 15 days, the mothers will receive mediterranean diet based on olive oil. Then, lactating women receive 30gr/day olive oil (standard group. Human milk will be collected during the first breastfeeding of the day (10 ml) at three times : Days 0 corresponding to the usual diet , at day 15 after the Mediterranean diet and at day 30, after the study diet.
  Arms: Olive oil

SUMMARY:
We propose to measure the LCPUFA human milk (linolenic acid, linoleic acid, docosahexaenoic acid, arachidonic acid) according to fatty acids nature and quantities consumed by lactating women

DETAILED DESCRIPTION:
n-3 and n-6 long chain polyunsaturated fatty acids (LCPUFA) are essential particularly to neurodevelopment of newborn infants. Many variations in essential PUFA and LCPUFA content of human milk are observed according to countries and dietary habits of the mothers.

Maternal diet supplementation of LCPUFA of lactating women may increase LCPUFA human milk according to consensus recommendations.

This clinical trial is performed to evaluate the effect of different of consumption of n-3 fatty acids (linolenic acid) in different forms (oils or margarine) in the human milk composition.

Each diet will last 30 days. During the first period of 15 days, the mothers will receive mediterranean diet based on olive oil. Then, lactating women will be randomised into four groups : one group will receive olive oil (standard group), one group supplemented in rapeseed oil, one group with n-3 margarine and one group with diet associating rapeseed oil and n-3 margarine.Human milk will be collected during the first breastfeeding of the day (10 ml) at three times : Days 0 corresponding to the usual diet , at day 15 after the Mediterranean diet and at day 30, after the study diet.

ELIGIBILITY:
Inclusion Criteria:

* Lactating women more than 1 month and less than 4 month with neonate whom term is between 37 and 42 gestational age
* Women who agree to consume fatty fish two times per week
* Free consent

Exclusion Criteria:

* Women with multiple infants
* Chronic treatments more than 8 days
* Women with treatment during supplementation period
* Women with maternal pathology not compatible with breastfeed

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 82 (Actual)
Dates: Start 2011-09; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Acide linolenic 18 :3 n-3 analysis measured at day 30, compared to day 15 | 30 days

SECONDARY OUTCOMES:
Analysis of linolenic acid and linoleic acid ratio | 30 days
Analysis of arachidonic acid, docosahexanoic acid and their ratio | 30 days
Comparison of fatty acid composition of human milk before and after supplementation | 30 days
Analysis of trans fatty acids according diets | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Paul PEREZ, MD, PhD, Study Chair — University Hospital Bordeaux (France)
Locations (4):
- France (4):
  - Lactarium Hôpital Pellegrin Enfants CHU Bordeaux, Bordeaux
  - Lactarium CHU La Croix Rousse Lyon Néonatologie et Réanimation Néonatale, Lyon
  - Lactarium CHU Montpellier Pédiatrie 2, Montpellier
  - Lactarium Institut de Puériculture de Paris et de Périnatalogie, Paris

REFERENCES:
- [Background] Lauritzen L, Hansen HS, Jorgensen MH, Michaelsen KF. The essentiality of long chain n-3 fatty acids in relation to development and function of the brain and retina. Prog Lipid Res. 2001 Jan-Mar;40(1-2):1-94. doi: 10.1016/s0163-7827(00)00017-5. No abstract available. PMID 11137568
- [Background] Sauerwald TU, Hachey DL, Jensen CL, Chen H, Anderson RE, Heird WC. Intermediates in endogenous synthesis of C22:6 omega 3 and C20:4 omega 6 by term and preterm infants. Pediatr Res. 1997 Feb;41(2):183-7. doi: 10.1203/00006450-199702000-00005. PMID 9029636
- [Background] Cunnane SC, Francescutti V, Brenna JT, Crawford MA. Breast-fed infants achieve a higher rate of brain and whole body docosahexaenoate accumulation than formula-fed infants not consuming dietary docosahexaenoate. Lipids. 2000 Jan;35(1):105-11. doi: 10.1007/s11745-000-0501-6. PMID 10695931
- [Background] Innis SM, Gilley J, Werker J. Are human milk long-chain polyunsaturated fatty acids related to visual and neural development in breast-fed term infants? J Pediatr. 2001 Oct;139(4):532-8. doi: 10.1067/mpd.2001.118429. PMID 11598600
- [Background] Jorgensen MH, Hernell O, Hughes E, Michaelsen KF. Is there a relation between docosahexaenoic acid concentration in mothers' milk and visual development in term infants? J Pediatr Gastroenterol Nutr. 2001 Mar;32(3):293-6. doi: 10.1097/00005176-200103000-00011. PMID 11345178
- [Background] Simmer K, Patole SK, Rao SC. Long-chain polyunsaturated fatty acid supplementation in infants born at term. Cochrane Database Syst Rev. 2008 Jan 23;(1):CD000376. doi: 10.1002/14651858.CD000376.pub2. PMID 18253974
- [Background] Uauy R, Hoffman DR, Mena P, Llanos A, Birch EE. Term infant studies of DHA and ARA supplementation on neurodevelopment: results of randomized controlled trials. J Pediatr. 2003 Oct;143(4 Suppl):S17-25. doi: 10.1067/s0022-3476(03)00398-6. PMID 14597910
- [Background] Hoffman DR, Birch EE, Castaneda YS, Fawcett SL, Wheaton DH, Birch DG, Uauy R. Visual function in breast-fed term infants weaned to formula with or without long-chain polyunsaturates at 4 to 6 months: a randomized clinical trial. J Pediatr. 2003 Jun;142(6):669-77. doi: 10.1067/mpd.2003.213. PMID 12838196
- [Background] SanGiovanni JP, Berkey CS, Dwyer JT, Colditz GA. Dietary essential fatty acids, long-chain polyunsaturated fatty acids, and visual resolution acuity in healthy fullterm infants: a systematic review. Early Hum Dev. 2000 Mar;57(3):165-88. doi: 10.1016/s0378-3782(00)00050-5. PMID 10742608
- [Background] Innis SM, Adamkin DH, Hall RT, Kalhan SC, Lair C, Lim M, Stevens DC, Twist PF, Diersen-Schade DA, Harris CL, Merkel KL, Hansen JW. Docosahexaenoic acid and arachidonic acid enhance growth with no adverse effects in preterm infants fed formula. J Pediatr. 2002 May;140(5):547-54. doi: 10.1067/mpd.2002.123282. PMID 12032520
- [Background] Jensen CL, Voigt RG, Prager TC, Zou YL, Fraley JK, Rozelle JC, Turcich MR, Llorente AM, Anderson RE, Heird WC. Effects of maternal docosahexaenoic acid intake on visual function and neurodevelopment in breastfed term infants. Am J Clin Nutr. 2005 Jul;82(1):125-32. doi: 10.1093/ajcn.82.1.125. PMID 16002810
- [Background] Helland IB, Smith L, Saarem K, Saugstad OD, Drevon CA. Maternal supplementation with very-long-chain n-3 fatty acids during pregnancy and lactation augments children's IQ at 4 years of age. Pediatrics. 2003 Jan;111(1):e39-44. doi: 10.1542/peds.111.1.e39. PMID 12509593
- [Background] Fidler N, Sauerwald T, Pohl A, Demmelmair H, Koletzko B. Docosahexaenoic acid transfer into human milk after dietary supplementation: a randomized clinical trial. J Lipid Res. 2000 Sep;41(9):1376-83. PMID 10974044
- [Background] Birch EE, Garfield S, Hoffman DR, Uauy R, Birch DG. A randomized controlled trial of early dietary supply of long-chain polyunsaturated fatty acids and mental development in term infants. Dev Med Child Neurol. 2000 Mar;42(3):174-81. doi: 10.1017/s0012162200000311. PMID 10755457
- [Background] Innis SM. Human milk: maternal dietary lipids and infant development. Proc Nutr Soc. 2007 Aug;66(3):397-404. doi: 10.1017/S0029665107005666. PMID 17637092
- [Background] Koletzko B, Lien E, Agostoni C, Bohles H, Campoy C, Cetin I, Decsi T, Dudenhausen JW, Dupont C, Forsyth S, Hoesli I, Holzgreve W, Lapillonne A, Putet G, Secher NJ, Symonds M, Szajewska H, Willatts P, Uauy R; World Association of Perinatal Medicine Dietary Guidelines Working Group. The roles of long-chain polyunsaturated fatty acids in pregnancy, lactation and infancy: review of current knowledge and consensus recommendations. J Perinat Med. 2008;36(1):5-14. doi: 10.1515/JPM.2008.001. PMID 18184094
- [Background] Yuhas R, Pramuk K, Lien EL. Human milk fatty acid composition from nine countries varies most in DHA. Lipids. 2006 Sep;41(9):851-8. doi: 10.1007/s11745-006-5040-7. PMID 17152922
- [Background] Gibson RA, Neumann MA, Makrides M. Effect of increasing breast milk docosahexaenoic acid on plasma and erythrocyte phospholipid fatty acids and neural indices of exclusively breast fed infants. Eur J Clin Nutr. 1997 Sep;51(9):578-84. doi: 10.1038/sj.ejcn.1600446. PMID 9306083
- [Background] Billeaud C, Bougle D, Sarda P, Combe N, Mazette S, Babin F, Entressangles B, Descomps B, Nouvelot A, Mendy F. Effects of preterm infant formula supplementation with alpha-linolenic acid with a linoleate/alpha-linolenate ratio of 6: a multicentric study. Eur J Clin Nutr. 1997 Aug;51(8):520-6. doi: 10.1038/sj.ejcn.1600436. PMID 11248877
- [Background] Francois CA, Connor SL, Wander RC, Connor WE. Acute effects of dietary fatty acids on the fatty acids of human milk. Am J Clin Nutr. 1998 Feb;67(2):301-8. doi: 10.1093/ajcn/67.2.301. PMID 9459379
- [Background] Molto-Puigmarti C, Castellote AI, Carbonell-Estrany X, Lopez-Sabater MC. Differences in fat content and fatty acid proportions among colostrum, transitional, and mature milk from women delivering very preterm, preterm, and term infants. Clin Nutr. 2011 Feb;30(1):116-23. doi: 10.1016/j.clnu.2010.07.013. Epub 2010 Aug 25. PMID 20800325